CLINICAL TRIAL: NCT01237015
Title: Effect of Nasal Continuous Positive Airway Pressure (CPAP) on Sucking, Swallowing and Coordination of Breathing and Swallowing During Oral Feeding in Human Neonates
Brief Title: Effect of Nasal Continuous Positive Airway Pressure (CPAP) on Oral Feeding in Human Neonates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Dre Céline Catelin, Centre Hospitalier Universitaire de Sherbrooke
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 07-157
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2010-11

CONDITIONS: Oral Feeding in Human Neonates During Nasal CPAP
Keywords: Neonate; Oral feeding; Nasal CPAP; Sucking; Swallowing; Breathing
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Infant Flow nasal CPAP — Infant Flow nasal CPAP 5 cm H2O

SUMMARY:
Current knowledge suggests that, to be successful, oral feeding in preterm babies should be initiated as soon as possible, often at an age where immature respiration still requires ventilatory support in the form of continuous positive airway pressure (CPAP). While some neonatologist teams claim great success with initiation of oral feeding in immature babies with CPAP, others strictly wait for CPAP to be no longer necessary before any attempt at oral feeding. Such controversy is fuelled by ignorance of the effects of CPAP on nutritive sucking and swallowing, including their coordination with breathing, and the fear to induce deleterious problems such as pulmonary aspiration of milk and/or respiratory failure. Ensuing delay in becoming proficient with oral feeding unduly prolongs hospital stays of preterm babies.

The aim of this study is to evaluate the effects of nasal CPAP on oral feeding in human neonates. More specifically, CPAP effects on nutritive sucking and swallowing, including on breathing-swallowing coordination, will be carefully assessed. The investigators hypothesize that nasal CPAP will lead to no or minimal alterations of breathing-nutritive swallowing coordination and will not induce deleterious cardiorespiratory events.

Accordingly, each neonate will be evaluated during 2 bottle feedings spaced of 24 h, one with nasal CPAP 5 cm H2O and the other without any CPAP. Sucking and swallowing activity, respiration, heart rate and oxygenation will be continuously recorded before, during and after bottle-feeding.

By filling a gap in knowledge, results from the study will hopefully help neonatologists afraid of doing more harm than good when initiating bottle-feeding in preterm babies under CPAP to join the many teams for whom it is no more a problem.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 24 weeks or more
* Hospitalized in the neonatology unit or the maternity unit of CHUS Fleurimont
* Feeds by complete oral feeding since 24 hours or more

Exclusion Criteria:

* Upper airways anomaly
* Brain injury : periventricular leukomalacia or intracranial hemorrhage > grade III (Papile classification)
* Neuromuscular disease
* Life-threatening congenital disease
* Any symptomatic intercurrent acute disease (ex.: infection)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Continuous monitoring of sucking, swallowing, breathing and cardiac parameters | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Praud, MD-PhD, Study Director — Centre de recherche clinique Étienne Lebel; Céline Catelin, MD, Study Director — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke - Fleurimont, Sherbrooke, Quebec, Canada